CLINICAL TRIAL: NCT03917238
Title: Comparison of the Beta Cell Mass During and Shortly After the Honeymoon Phase of Type 1 Diabetes Using Gallium-68-exendin PET
Brief Title: Beta Cell Imaging During and Shortly After the Honeymoon Phase of T1D
Acronym: Honeymoon
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL61915.091.17
Record Dates: First submitted 2019-03-13; First posted 2019-04-17 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with T1D (Other): gallium-68-exendin followed by a PET/CT scan (twice)
  Interventions: Radiation: gallium-68-exendin injection followed by PET/CT scan

INTERVENTIONS:
Radiation: gallium-68-exendin injection followed by PET/CT scan — After injecting gallium-68-exendin, a PET/CT scan is performed during the honeymoon phase and repeated once the honeymoon phase has ended

SUMMARY:
The primary goal is to correlate beta cell mass to beta cell function from measurements during and shortly after the honeymoon phase of type 1 diabetes, to improve understanding of the change in metabolic control after the honeymoon phase.

DETAILED DESCRIPTION:
The exact role of beta cell mass during the development and course of diabetes is still poorly understood. Further research on beta cell mass is essential to obtain more insights that might aid in the development of diabetes treatment. This study aims at a specific phase of T1D that is called the 'honeymoon phase' or period of partial remission. Once insulin treatment has started, the honeymoon phase will arise in most patients. In this period, T1D patients become temporarily less insulin-dependent. Unfortunately, the honeymoon phase is only temporary, in which a decline in blood glucose regulation will be seen afterwards, leading to an increasing demand for insulin. To increase understanding of this change in metabolic control after the honeymoon phase, repeated measurements of the beta cell mass and function are performed during and shortly after the honeymoon phase. The comparison of both measurements might lead to an increased understanding whether changes in insulin demand after the honeymoon phase is mainly dependent on a decline in the beta cell mass, or because of a decrease in functional beta cells. The outcome of this study can provide new insights, which can contribute to the development of novel treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 16 years
* Diagnosed with T1D
* Presence of anti-GAD
* Subject is in honeymoon phase
* 17 ≤ BMI ≥ 30 kg/m^2 at moment of visit
* Ability to sign informed consent

Exclusion Criteria:

* Previous treatment (within 6 months) with synthetic Exendin (Exenatide, Byetta®) or Dipeptidyl-Peptidase IV inhibitors
* Liver disease
* Renal disease
* Pregnancy or the wish to become pregnant within 6 months after the study
* Breastfeeding
* BMI <17 kg/m2 or BMI >30 kg/m2
* Age <16 years
* When the end of the honeymoon phase is not observed within 11 to 13 months after the inclusion of the subject
* Inability to sign informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2019-10-11 (Actual); Primary Completion 2026-11-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Pancreatic uptake of gallium-68-NODAGA-exendin-4 | 2 years
  Pancreatic uptake is measured by quantitative analysis of PET/CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Martin Gotthardt, Prof. Dr., Principal Investigator — Radiology and Nuclear Medicine, Radboudumc, Nijmegen, The Netherlands
Locations (2):
- Netherlands (2):
  - Radboud university medical center, Nijmegen, Gelderland
  - Diabeter, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: No